CLINICAL TRIAL: NCT01552928
Title: A Phase 1, Randomized, Double-blind, Placebo- and Positive-controlled, 4-Period Crossover Trial to Assess the Effect of Anagrelide Hydrochloride on QT/QTc Interval in Healthy Men and Women.
Brief Title: Effect of Anagrelide Hydrochloride on Any Changes in Heart Function in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD422-111; 2011-005288-26 (EudraCT Number)
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — anagrelide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Anagrelide Therapeutic (0.5 mg) (Experimental)
  Interventions: Drug: Anagrelide 0.5 mg
- Anagrelide Supratherapeutic (2.5 mg) (Experimental)
  Interventions: Drug: Anagrelide 2.5 mg
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anagrelide 0.5 mg — 0.5mg Anagrelide single oral dose
  Other Names: Agrylin, Xagrid
  Arms: Anagrelide Therapeutic (0.5 mg)
Drug: Anagrelide 2.5 mg — 2.5mg Anagrelide single oral dose
  Arms: Anagrelide Supratherapeutic (2.5 mg)
Drug: Moxifloxacin — 400 mg Moxifloxacin single oral dose
  Arms: Moxifloxacin
Drug: Placebo — Anagrelide placebo + Moxifloxacin placebo single oral dose
  Arms: Placebo

SUMMARY:
According to the ICH Guidance Document E14, all non-antiarrhythmic drugs should be evaluated for their ability to prolong the QT interval which represents the duration of ventricular depolarization and subsequent repolarization. The primary objective of the study is to assess the effect of anagrelide on QT/QTc interval following a therapeutic and supratherapeutic dose of anagrelide when compared to placebo and a positive control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the screening period. This inclusion criteria will only be assessed at the screening visit.
* Subject is willing to comply with any applicable contraceptive requirements of the protocol and is: male, or non-pregnant non lactating female, or females must be at least 90 days post-partum or nulliparous.
* Satisfactory medical assessment with no clinically or relevant abnormalities in medical history, physical examination, vital signs, ECG, and clinical laboratory evaluation as assessed by the investigator.

Exclusion Criteria:

* Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or could affect clinical or laboratory assessments.

  a- Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Significant illness, as judged by the Investigator, within 2 weeks of the first dose of investigational product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2012-07-25 (Actual); Study Completion 2012-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Biotrial, Rueil-Malmaison, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg: A single oral dose of 0.5 mg of anagrelide on Day 1 for Period 1; then a single oral dose of 2.5 mg of anagrelide on Day 1 for Period 2; then a single oral dose of placebo on Day 1 for Period 3; then a single oral dose of 400 mg of moxifloxacin on Day 1 for Period 4.
- Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo: A single oral dose of 2.5 mg of anagrelide on Day 1 for Period 1; then a single oral dose of 400 mg of moxifloxacin on Day 1 for Period 2; then a single oral dose of 0.5 mg of anagrelide on Day 1 for Period 3; then a single oral dose of placebo on Day 1 for Period 4.
- Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg: A single oral dose of 400 mg of moxifloxacin on Day 1 for Period 1; then a single oral dose of placebo on Day 1 for Period 2; then a single oral dose of 2.5 mg of anagrelide on Day 1 for Period 3; then a single oral dose of 0.5 mg of anagrelide on Day 1 for Period 4.
- Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg: A single oral dose of placebo on Day 1 for Period 1; then a single oral dose of 0.5 mg of anagrelide on Day 1 for Period 2; then a single oral dose of 400 mg of moxifloxacin on Day 1 for Period 3; then a single oral dose of 2.5 mg of anagrelide on Day 1 for Period 4.
Period: Period 1
Arm/Group | Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg | Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo | Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg | Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg
Started | 14 | 15 | 15 | 16
Completed | 14 | 15 | 15 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg | Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo | Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg | Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg
Started | 14 | 15 | 15 | 16
Completed | 14 | 15 | 15 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg | Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo | Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg | Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg
Started | 14 | 15 | 15 | 16
Completed | 14 | 15 | 14 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period 4
Arm/Group | Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg | Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo | Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg | Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg
Started | 14 | 15 | 14 | 16
Completed | 14 | 15 | 14 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anag 0.5 mg, Then Anag 2.5 mg, Then Placebo, Then Mox 400 mg | Anag 2.5 mg, Then Mox 400 mg, Then Anag 0.5 mg, Then Placebo | Mox 400 mg, Then Placebo, Then Anag 2.5 mg, Then Anag 0.5 mg | Placebo, Then Anag 0.5 mg, Then Mox 400 mg, Then Anag 2.5 mg | Total
Number analyzed (Participants) | 14 | 15 | 15 | 16 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 15 | 16 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.1 (6.44) | 28.4 (7.7) | 29.5 (5.83) | 30.4 (8.02) | 29.2 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 7 | 25
  Male | 8 | 9 | 9 | 9 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  FRANCE | 14 | 15 | 15 | 16 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcNi Intervals at Subject-Specific Time of Maximum Plasma Concentration (Tmax)
Description: QT interval corrected for heart rate using the subject-specific method (QTcNi) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value.
Time Frame: Over 12 hours post-dose
Population: Full Analysis Set (FAS) consists of subjects in the Safety Analysis Set who had at least 1 electrocardiogram (ECG). Safety Analysis Set consists of subjects who received at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Anagrelide 0.5 mg: A single oral dose of 0.5 mg of anagrelide
- Anagrelide 2.5 mg: A single oral dose of 2.5 mg of anagrelide
- Moxifloxacin 400 mg: A single oral dose of 400 mg of moxifloxacin
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 51 | 55 | 55
msec | 4.4 [2.0 to 6.8] | 8.2 [4.9 to 11.6] | 11.3 [9.0 to 13.7]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.004, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Mean Difference Changes From Baseline Versus Placebo in Heart Rate at Subject-Specific Tmax
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 51 | 55 | 55
beats per minute | 4.5 [2.7 to 6.2] | 21.8 [18.3 to 25.4] | 2.9 [1.5 to 4.3]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.001, ANCOVA

3. Secondary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcF Intervals at Subject-Specific Tmax
Description: QT interval corrected for heart rate using Fridericia's method (QTcF) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 51 | 55 | 55
msec | 3.7 [1.3 to 6.1] | 4.5 [0.8 to 8.1] | 10.8 [8.5 to 13.1]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p = 0.044, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcB Intervals at Subject-Specific Tmax
Description: QT interval corrected for heart rate using Bazett's method (QTcB) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 51 | 55 | 55
msec | 8.5 [4.9 to 12.0] | 25.5 [20.3 to 30.6] | 14.0 [11.0 to 17.1]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Mean Difference Changes From Baseline Versus Placebo in QT Intervals at Subject-Specific Tmax
Description: The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 51 | 55 | 55
msec | -6.1 [-9.5 to -2.8] | -34.3 [-40.5 to -28.1] | 4.3 [0.8 to 7.7]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.003, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.043, ANCOVA

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of 0.5 mg Anagrelide in Males and Females
Time Frame: Over 12 hours post-dose
Population: Pharmacokinetic Analysis Set consists of all subjects in the Safety Analysis Set who had evaluable concentration-time profiles for anagrelide, BCH24426, or moxifloxacin.
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- Anagrelide 0.5 mg (Males); Anagrelide 0.5 mg (Females): A single oral dose of 0.5 mg of anagrelide
Arm/Group | Anagrelide 0.5 mg (Males) | Anagrelide 0.5 mg (Females)
Number analyzed (Participants) | 34 | 25
ng/ml | 2.083 (0.975) | 3.64 (1.959)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of 2.5 mg Anagrelide in Males and Females
Time Frame: Over 12 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- Anagrelide 2.5mg (Males); Anagrelide 2.5mg (Females): A single oral dose of 2.5 mg of anagrelide
Arm/Group | Anagrelide 2.5mg (Males) | Anagrelide 2.5mg (Females)
Number analyzed (Participants) | 35 | 25
ng/ml | 10.592 (4.871) | 16.378 (10.224)

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Metabolite of 0.5 mg Anagrelide (BCH24426) in Males and Females
Time Frame: Over 12 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- BCH24426 (Males); BCH24426 (Females): Metabolite from a single oral dose of 0.5 mg of anagrelide
Arm/Group | BCH24426 (Males) | BCH24426 (Females)
Number analyzed (Participants) | 34 | 25
ng/ml | 3.731 (1.257) | 4.534 (1.405)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Metabolite of 2.5 mg Anagrelide (BCH24426) in Males and Females
Time Frame: Over 12 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- BCH24426 (Males); BCH24426 (Females): Metabolite from a single oral dose of 2.5 mg of anagrelide
Arm/Group | BCH24426 (Males) | BCH24426 (Females)
Number analyzed (Participants) | 35 | 25
ng/ml | 18.927 (6.016) | 23.785 (7.952)

10. Primary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcNi Intervals From Time-Matched Analysis by Largest Time Point
Description: QT interval corrected for heart rate using the subject-specific method (QTcNi) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value. The largest time point refers to the estimated largest mean difference between each treatment and placebo among all time points. Values for different treatments can come from different time points.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 50 | 55 | 53
msec | 7.0 [4.2 to 9.8] | 13.0 [10.3 to 15.7] | 12.6 [9.9 to 15.2]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

11. Primary Outcome: Mean Difference Changes From Baseline Versus Placebo in Heart Rate From Time-Matched Analysis by Largest Time Point
Description: The largest time point refers to the estimated largest mean difference between each treatment and placebo among all time points. Values for different treatments can come from different time points.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 50 | 54 | 53
beats per minute | 7.8 [5.3 to 10.4] | 29.1 [26.6 to 31.6] | 4.3 [1.8 to 6.7]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.004, ANCOVA

12. Primary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcF Intervals From Time-Matched Analysis by Largest Time Point
Description: QT interval corrected for heart rate using Fridericia's method (QTcF) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value. The largest time point refers to the estimated largest mean difference between each treatment and placebo among all time points. Values for different treatments can come from different time points.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 50 | 55 | 53
msec | 5.0 [2.1 to 8.0] | 10.0 [7.3 to 12.7] | 11.8 [8.9 to 14.8]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.005, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

13. Primary Outcome: Mean Difference Changes From Baseline Versus Placebo in QTcB Intervals From Time-Matched Analysis by Largest Time Point
Description: QT interval corrected for heart rate using Bazett's method (QTcB) at the subject-specific time of maximum plasma concentration. The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value. The largest time point refers to the estimated largest mean difference between each treatment and placebo among all time points. Values for different treatments can come from different time points.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 50 | 56 | 55
msec | -2.9 [-5.6 to -0.2] | -18.1 [-20.7 to -15.4] | -2.3 [-5.0 to 0.4]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.078, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p = 0.156, ANCOVA

14. Primary Outcome: Mean Difference Changes From Baseline Versus Placebo in QT Intervals From Time-Matched Analysis by Largest Time Point
Description: The QT interval is the time it takes for the ventricles of the heart to contract and relax. Data were subtracted from the placebo value. The largest time point refers to the estimated largest mean difference between each treatment and placebo among all time points. Values for different treatments can come from different time points.
Time Frame: Over 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Anagrelide 0.5 mg | Anagrelide 2.5 mg | Moxifloxacin 400 mg
Number analyzed (Participants) | 49 | 54 | 56
msec | 1.7 [-2.0 to 5.4] | -2.4 [-6.0 to 1.2] | 9.6 [5.2 to 14.1]
Statistical Analysis 1: Comparison: Anagrelide 0.5 mg; Test type: Superiority or Other; p = 0.439, ANCOVA
Statistical Analysis 2: Comparison: Anagrelide 2.5 mg; Test type: Superiority or Other; p = 0.274, ANCOVA
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | Anagrelide 0.5mg | Anagrelide 2.5mg | Moxifloxacin 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 13/59 | 49/60 | 2/60 | 0/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide 0.5mg (N=59) | Anagrelide 2.5mg (N=60) | Moxifloxacin 400mg (N=60) | Placebo (N=60)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 17 (17) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 14 (14) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 44 (44) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.